CLINICAL TRIAL: NCT05931835
Title: Luma Vision's Feasibility Study on the VERAFEYE System
Brief Title: Feasibility Study on the VERAFEYE System
Acronym: LUMINIzE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LUMA Vision Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LUMINIzE-P001
Record Dates: First submitted 2023-06-09; First posted 2023-07-05 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Atrial Septal Defect; Atrial Fibrillation; Atrial Arrhythmia; Left Atrial Appendage Closure
MeSH Terms: conditions — Heart Septal Defects, Atrial; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Catheter-ablation and closure procedures arm (Experimental): Subjects entitled to undergo a catheter-based ablation treatment for typical atrial flutter or atrial fibrillation and subjects entitled to undergo a left atrial appendage/atrial septal defect closure procedure
  Interventions: Device: VERAFEYE System

INTERVENTIONS:
Device: VERAFEYE System — The VERAFEYE System will be used during standard of care, catheter-based treatments for atrial flutter or atrial fibrillation; or left atrial appendage/atrial septal defect closure procedures.

SUMMARY:
The objective of the study is to evaluate the performance of the VERAFEYE System in subjects entitled to undergo a standard of care ablation or closure procedure.

Results from this study will be used to guide development and refinement the VERAFEYE System. The study is not designed to collect data for product approval and as such does not have a safety or efficacy endpoint.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject is 18 to 80 years of age at the time of consent
* Subject is scheduled to undergo a standard of care, de-novo catheter-ablation procedure to treat typical AFL or AF; or left atrial appendage (LAA)/ atrial septal defect (ASD) closure procedure
* Subject is able to understand and willing to provide written informed consent

Key Exclusion Criteria:

* Any of the following within 6 months prior to enrolment:

  * Cardiac surgery including coronary artery bypass grafting, ventriculotomy, atriotomy
  * Thromboembolic event (stroke), transient ischemic attack (TIA) or neurological disturbances
  * Myocardial infarction
  * Any surgical or percutaneous cardiac procedure including coronary intervention and cardiac ablation
  * Dilated or hypertropic cardiomyopathy
* Any planned surgical or endovascular intervention within 30 days before or after the ablation, or LAA/ASD closure procedure.
* Any of the following cardiac conditions:

  * New York Heart Association (NYHA) class IV
  * Left ventricular ejection fraction (LVEF) < 30%
  * Implanted with a cardiac rhythm management device (pacemaker, CRT, ICD, loop recorder)
  * Presence of intramural thrombus, tumor, or other abnormality that precludes vascular access, catheter introduction, or manipulation
  * Active coronary ischemia, significant valvular heart disease, or hemodynamically significant congenital cardiac abnormality
* Body mass index (BMI) > 40 kg/m2
* Body weight < 50kg
* Pregnant women or women who plan to become pregnant during the course of their participation in the study (women should either be of non- childbearing potential at the time of enrolment (as documented in the medical file) or have a negative pregnancy test within the previous 7 days prior to the ablation, or LAA/ASD closure procedure)
* Life expectancy less than 12 months
* Subjects who are currently enrolled in another study
* Subjects with a thrombus or pericardial effusion detected in the LA/LAA during standard of care imaging

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mater Private Network, Dublin, Leinster, Ireland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 18 enrolled participants, 17 underwent catheter ablation procedure with VERAFEYE System.
Pre-assignment Details: 1 of 18 enrolled subjects was classified as an intent subject (no VERAFEYE Imaging Catheter inserted into the body).
Groups:
- Catheter-ablation Arm: Subjects entitled to undergo a catheter-based ablation treatment for typical atrial flutter or atrial fibrillation.
Period: Overall Study
Arm/Group | Catheter-ablation Arm
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Procedure subjects
Arm/Group | Catheter-ablation Arm
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Ireland | 17
Height [Mean (Standard Deviation); unit: cm] | 176.9 (11.6)
Weight [Mean (Standard Deviation); unit: kg] | 91.2 (15.7)
Resting Heart Rate [Mean (Standard Deviation); unit: bpm] | 75.8 (18.7)
Systolic BP [Mean (Standard Deviation); unit: mmHg] | 135.4 (21.1)
Diastolic BP [Mean (Standard Deviation); unit: mmHg] | 85.6 (13.8)
12-lead ECG at Baseline [Count of Participants; unit: Participants]
  Atrial Fibrillation | 7
  Sinus Rhythm | 7
  Atrial Flutter | 2
  Atrial Fibrillation AND Atrial Flutter | 1

OUTCOME MEASURES:

1. Primary Outcome: Physician Feedback on VERAFEYE System
Description: The objective of the study is to collect physician feedback by means of a questionnaire on the VERAFEYE System. Results from this study may be used to guide development and refinement of the VERAFEYE System.
Time Frame: During the procedure (up to two hours)
Measure: Number; unit: percentage of participants
Arm/Group | Catheter-ablation Arm
Number analyzed (Participants) | 17
percentage of participants
  VERAFEYE Imaging Catheter (VIC) rated as able to navigate to RA | 100
  Introduction of the VIC into the vasculature&navigation to the RA rated as acceptable and above | 100
  Visualization of major anatomical structures (excl. LA) from the RA rated as acceptable and above | 100
  Visualization of the LA from the RA rated acceptable and above | 100
  Articulation/maneuverability of the VIC rated acceptable and above | 100
  Ability of the System to visualize the third party devices rated acceptable and above | 100
  Overall image quality 2D rated acceptable and above | 94.1
  Overall image quality 4D rated acceptable and above | 88.2
  No anatomical locations were difficult to reach with the VIC | 100
  How feasible was it for you to integrate the usage of the System into your workflow? rated as easy | 100
  Were the views and the possibilities for manipulating the views helpful? slightly helpful and above | 100

ADVERSE EVENTS:
Time Frame: 7 days post index procedure
Description: No adverse events reported
Arm/Group | Catheter-ablation Arm
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

LIMITATIONS AND CAVEATS:
LUMINIzE was designed as a single-center feasibility study without safety/effectiveness endpoints since the study was intended to collect data for future R&D development. High volume ablating center with experienced Investigators was selected for participation in this study. Therefore, the procedural data reported in this clinical study may be different in other settings as it is expected that operator experience can positively influence the outcomes of the procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT05931835/Prot_SAP_000.pdf